CLINICAL TRIAL: NCT04943523
Title: Effects of Krill Oil Supplementation on Muscle Mass and Function in People With Muscle Weakness and Type 2 Diabetes
Brief Title: Krill Oil and Muscle Weakness in Type 2 Diabetes
Acronym: KRIMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA HM-2021-010
Record Dates: First submitted 2021-06-22; First posted 2021-06-29 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Plant Oils

STUDY DESIGN:
Intervention Model Description: Parallel Group Randomised Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): vegetable oil 4g/day
  Interventions: Dietary Supplement: Vegetable Oil
- Krill Oil (Active Comparator): Krill Oil 4g/day
  Interventions: Dietary Supplement: Krill Oil

INTERVENTIONS:
Dietary Supplement: Krill Oil — Krill oil supplements 4g/day
  Arms: Krill Oil
Dietary Supplement: Vegetable Oil — vegetable oil supplements 4g/day
  Arms: Placebo

SUMMARY:
The age-related loss of muscle mass and function, sarcopenia, has several deleterious effects, such as a reduction in the quality of life and an increase in the incidence of falls, often leading to hospitalisation. The prevalence of sarcopenia is unclear but is estimated to be between 4.6 and 7.9% and the loss of skeletal muscle mass and function is accelerated in people with type 2 diabetes. With the percentage of older people and the percentage of people with type 2 diabetes predicted to rise in coming years it is crucial to develop therapies to increase muscle mass and function. Alterations in nutrition have also been suggested to be of therapeutic use in sarcopenia. Epidemiological data showed that the consumption of fatty fish is positively associated with muscle function in older population, indicating a potential role for long-chain n-3 polyunsaturated fatty acids (LCn-3 PUFA) in increasing muscle mass and function in older people. The aim of the current study, therefore, is to determine the effects of krill oil supplementation on muscle size and function in adults with muscle weakness and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Physician confirmed type 2 diabetes.
* Age >/= 40 years
* No changes in anti-diabetic medication in the last 3 months.
* Muscle weakness (grip strength <27kg and females <16kg)

Exclusion Criteria:

* BMI of 45 or higher
* BP of 160/100mmHg or higher
* Cancer or cancer that has been in remission <5 years
* Any medical condition that prevents participants from exercising safely
* On anticoagulant therapy
* Allergies to seafood
* Regular consumption of more than 2 portions of oily fish per week
* Currently consuming omega-3 supplements

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Grip strength | Change from baseline to one year
  Change in Grip strength

SECONDARY OUTCOMES:
SPPB | Change from baseline to one year
  Change in Short performance physical battery test
HbA1c | Change from baseline to one year
  Change in glycated haemoglobin
Blood pressure | Change from baseline to one year
  Change in blood pressure
body mass | Change from baseline to one year
  Change in body mass
Lean mass | Change from baseline to one year
  Change in lean mass
Body fat | Change from baseline to one year
  Change in body fat
BMC | Change from baseline to one year
  Change in bone mineral content
BMD | Change from baseline to one year
  Change in bone mineral density
Erythrocyte fatty acid profile | Change from baseline to one year
  Change in Erythrocyte fatty acid profile

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa AlOzairi, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait